CLINICAL TRIAL: NCT07275515
Title: DIROXIMEL FUMARATE TO REDUCE PERIHAEMATOMAL OEDEMA IN INTRACEREBRAL HAEMORRHAGE: A DOUBLE BLIND RANDOMIZED CLINICAL TRIAL (DARLENE)
Brief Title: DIROXIMEL FUMARATE TO REDUCE PERIHAEMATOMAL OEDEMA IN INTRACEREBRAL HAEMORRHAGE: DOUBLE BLIND RANDOMIZED CLINICAL TRIAL
Acronym: DARLENE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministère de la Santé (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024_0474; 2025-522687-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: proof of concept; multicenter; stroke; randomization; double-blind, placebo-controlled; France; DRF group VS Placebo group
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacist, CRA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DRF group (Experimental): 2*231 mg of Diroximel Fumarate (DRF) per day for 7 days then 4*231 mg per day for 14 days.
  Interventions: Drug: DRF
- Placebo group (Placebo Comparator): 2 capsules of matching placebo per day for 7 days than 4 capsules of matching placebo per day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DRF — 2*231 mg of Diroximel Fumarate (DRF) per day for 7 days then 4*231 mg per day for 14 days.
  Arms: DRF group
Drug: Placebo — 2 capsules of matching placebo per day for 7 days than 4 capsules of matching placebo per day for 14 days.
  Arms: Placebo group

SUMMARY:
Spontaneous intracerebral haemorrhage (ICH) is a life-threatening condition, still devoided of specific treatment. Peri-haematomal oedema (PHO) develops in the ensuing days after ICH onset and worsens functional outcome. Hence, PHO is a promising therapeutic target but until now there is no specific treatment for PHO. The occurrence and growth of PHO is mainly mediated by inflammation. We hypothesize that a modulation of inflammation is effective in reducing PHO growth, therefore improving the functional outcome of ICH patients. From animal studies to human post-mortem studies, our team has demonstrated a key role for erythroid-related nuclear factor 2 (Nrf2) in PHO. Indeed, this transcription factor promotes the protective effect of inflammation: Nrf2 activation enhances antioxidant defenses and increases rates of blood resorption. Therefore, Nrf2 emerges as a promising and innovative therapeutic target. Taking into account the prolonged time interval between de novo drug discovery and use in clinical practice, drug repurposing is an interesting option for the unmet clinical need of reducing PHO. We chose Diroximel Fumarate (DRF) which is a safe and effective Nrf2 activator widely used in multiple sclerosis (dimethyl fumarate is on the market since 2013, and DRF since 2019) to modulate inflammation and to establish the efficacy of Nrf2 activation in reducing PHO growth and, ultimately, in improving the functional prognosis after ICH.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older (no upper age limit)
2. Patients admitted for a first-ever or recurrent (occurred more than 1 year before) symptomatic supratentorial spontaneous ICH confirmed by brain imaging
3. Administration of study treatment no later than 48 hours after symptom onset or since last seen normal
4. Written consent obtained
5. Patient with social insurance in France
6. Patient willing to comply with all study procedures and duration

Exclusion Criteria:

1. Massive ICH for Investigational medicinal product seems futile (hematoma volume is estimated > 60ml)
2. Severe coma (Glasgow Coma Scale <6)
3. Pure intraventricular hemorrhage
4. ICH suspected to result from a preceding trauma, an identified intracranial vascular malformation, venous thrombosis, tumor or hemorrhagic transformation within an infarct
5. Patient planned for surgical evacuation of ICH before randomization (Evacuation, Decompressive hemicraniectomy, External ventricular drain)
6. Patient with a known indication for DRF treatment (e.g. multiple sclerosis) or any other NrF2 agonist (dimethyl fumarate; Tecfidera)
7. Patient with contraindication to DRF: patients with known hypersensitivity to DRF, or to any of the excipients of VUMERITY (patients taking dimethyl fumarate)
8. Severe lymphopenia at admission (lymphocyte counts < 0.5 x 109/L)
9. Medical history of progressive multifocal leukoencephalopathy
10. Severe swallowing disorder and/or nasogastric tube required
11. Severe pre-ICH dependency (modified Rankin score of 5)
12. Life expectancy < 1 year related to comorbidities
13. Late-stage organ (acute cardiac, renal or hepatic failure)
14. Decision already taken for palliative (end of life) care with withdrawal of active treatment
15. Pregnancy or breastfeeding or Women of childbearing age without effective contraception (a pregnancy test will be done)
16. Adults who are deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Absolute volume of PHO assessed at 8 ± 1 days with brain non-contrast CT (NCCT) scan. | at 8 ± 1 days

SECONDARY OUTCOMES:
Functional outcome: global disability assessed by overall distribution of mRS score at 6 months (end of follow-up) (shift analysis) | at 6 months
The rate of severe adverse events occurring between the date of randomization and the end of follow-up (six-month visit). | At 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided